CLINICAL TRIAL: NCT01353209
Title: Trial of Letrozole in Lymphangioleiomyomatosis
Brief Title: Letrozole for Lymphangioleiomyomatosis
Acronym: TRAIL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Francis McCormack, Professor and Director, Pulmonary, Critical Care and Sleep Medicine, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5708
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Lymphangioleiomyomatosis
Keywords: Lymphangiomyomatosis; Postmenopausal
MeSH Terms: conditions — Lymphangioleiomyomatosis | interventions — Letrozole; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Letrozole (Experimental): Patients are placed on letrozole, 1 tablet (2.5 mg) daily for one year
  Interventions: Drug: Letrozole
- Placebo (Placebo Comparator): Patients are placed on placebo, 1 tablet daily for one year
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Letrozole — 2.5 mg daily for twelve months
  Other Names: Femara
  Arms: Letrozole
Drug: Placebo — placebo given daily for twelve months
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The hypothesis in this study is that estrogen suppression by an aromatase inhibitor in postmenopausal women with lymphangioleiomyomatosis (LAM) will prevent or delay progression of lung disease and result in a decrease in the rate of decline in FEV1

DETAILED DESCRIPTION:
Lymphangioleiomyomatosis, or LAM, is an uncommon, progressive, cystic lung disease that predominantly affects young women. Pulmonary parenchymal changes consistent with LAM are found in about one third of women with tuberous sclerosis complex (TSC), an autosomal dominant tumor suppressor syndrome. LAM also occurs in a sporadic form that is not associated with germline mutations in TSC genes. Recent evidence that recurrent LAM after lung transplantation results from seeding of the graft from a remote source and suggests a metastatic mechanism for the disease.

Since LAM occurs almost exclusively in women, and is exacerbated by pregnancy, menses and hormonal therapies suggest that estrogen suppression might be expected to prevent or delay progression of disease.

In postmenopausal women, estrogens are mainly derived from the action of the aromatase enzyme, which converts adrenal androgens (primarily androstenedione and testosterone) to estrone and estradiol. The suppression of estrogen biosynthesis in peripheral tissues can therefore be achieved by specifically inhibiting the aromatase enzyme. Letrozole is a nonsteroidal aromatase inhibitor (inhibitor of estrogen synthesis) that has been shown to be effective in other neoplasms that affect women, such as breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of based on compatible chest CT and at least one of the following:

  1. biopsy or cytology consistent with LAM, or
  2. tuberous sclerosis, renal angiomyolipoma, cystic abdominal lymphangiomas, or chylous effusion in the chest or abdomen, or
  3. serum VEGF-D ≥ 800 pg/uL.
* post bronchodilator FEV1 ≤80% predicted or DLCO ≤70% predicted or RV≥120% predicted
* female and postmenopausal status as defined by one of the following:

  1. prior bilateral oophorectomy or bilateral ovarian irradiation, or
  2. age greater than 55 years, and no menstrual period for 12 months or longer.
  3. age 18-55 years and estradiol level in the postmenopausal range in the absence of current use of progestational agents.

     * If still premenopausal, may enter if rendered medically postmenopausal on clinical grounds with the use of gonadotropin releasing hormone (e.g. leuprolide), as long as serum estradiol, FSH, and LH are in the postmenopausal range
* Patients with osteopenia or osteoporosis must be receiving appropriate treatment for their osteoporosis or osteopenia at entry into this study.

Exclusion Criteria:

* Known allergy to letrozole
* Inability to comply with pulmonary function tests or follow up visits.
* Treatment with investigational agents within 30 days
* Hormonal therapy (e.g. estrogen, progestin, LHRH agonists or antagonists, estrogen receptor blockers, estrogen receptor down regulators, aromatase inhibitors) within 30 days month of registration
* Medical or psychiatric conditions that would interfere with the ability to provide informed consent.
* abnormal hematologic and hepatic function as defined by the following at the time of randomization.:
* Neutrophils < 1500/mm3 and platelets < 100,000/mm3
* Bilirubin < 1.25 X upper limit of normal
* SGPT (ALT) or SGOT (AST) >2.5 X upper limit of normal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis X McCormack, MD, Principal Investigator — University of Cincinnati
Locations (9):
- United States (9):
  - Stanford University Medical Center, Stanford, California
  - Mayo Clinic, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Minor and James, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Deidentified demographics and outcomes can be shared. Because LAM is a rare disease, demographics will be limited. A data transfer agreement will be implemented between the University of Cincinnati and the requesting entity.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: immediately, indefinitely
Access Criteria: Email the PI: mccormfx@ucmail.uc.edu

REFERENCES:
- [Result] Lu C, Lee HS, Pappas GP, Dilling DF, Burger CD, Shifren A, Veeraraghavan S, Chapman JT, Parambil J, Ruoss SJ, Young LR, Hammes SR, Kopras EJ, Roads T, Krischer JP, McCormack FX; Trial of an Aromatase Inhibitor in Lymphangioleiomyomatosis Group. A Phase II Clinical Trial of an Aromatase Inhibitor for Postmenopausal Women with Lymphangioleiomyomatosis. Ann Am Thorac Soc. 2017 Jun;14(6):919-928. doi: 10.1513/AnnalsATS.201610-824OC. PMID 28570161

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were eligible for inclusion in the study if they were postmenopausal women with a definite diagnosis of pulmonary LAM and abnormal pulmonary function. Patients on sirolimus were required to wait three months before beginning this trial.
Groups:
- Placebo: Placebo: sugar pill given daily for twelve months
Period: Overall Study
Arm/Group | Letrozole | Placebo
Started | 9 | 8
Completed | 8 | 7
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Letrozole | Placebo | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 1 | 1 | 2
Age, Continuous [Median (Full Range); unit: years] | 57 [48 to 71] | 59 [44 to 68] | 58 [44 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 17
LAM subtyped [Number; unit: participants]
  Sporadic LAM | 6 | 8 | 14
  TSC LAM | 3 | 0 | 3
Sirolimus status [Count of Participants; unit: Participants]
  On sirolimus | 5 | 5 | 10
  Not on sirolimus | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Rate of Change in Forced Expiratory Volume in 1 Second in ml/Month
Description: FEV1 values reported are in liters or milliliters. There are no definite minimum and maximum values of FEV1 as it is a physiological measure of lung function and varies from individual to individual. Higher FEV1 scores indicate better lung function.
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: milliliters per month
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 8 | 7
milliliters per month | 1.04 [0.56 to 2.02] | 1.66 [0.77 to 2.63]
Statistical Analysis 1: Comparison: Letrozole vs Placebo; Test type: Superiority; p = 0.4, Mixed Models Analysis; Linear Mixed-Effects Model Adjusted for Sirolimus Use

2. Secondary Outcome: Post-bronchodilator FVC
Description: Post-bronchodilator FVC in milliliters
Time Frame: twelve months
Measure: Median (Full Range); unit: milliliters per month
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 8 | 7
milliliters per month | 2.58 [2.07 to 3.44] | 2.46 [1.26 to 3.21]
Statistical Analysis 1: Comparison: Letrozole vs Placebo; Test type: Superiority; p = 0.7, Mixed Models Analysis; Linear Mixed-Effects Model Adjusted for Sirolimus Use

3. Secondary Outcome: St George Respiratory Questionnaire
Description: Quality of Life scale for respiratory symptoms. This is a disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Scores range from 0 to 100, with higher scores indicating worse quality of life.
Time Frame: twelve months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 8 | 7
score on a scale | 38 [27 to 53] | 62 [38 to 82]
Statistical Analysis 1: Comparison: Letrozole vs Placebo; Test type: Superiority; p = 0.8, Regression, Linear; Linear Mixed-Effects Model Adjusted for Sirolimus Use
Statistical Analysis 2: Comparison: Letrozole vs Placebo; Test type: Superiority; p = .8, Regression, Linear

4. Secondary Outcome: Serum VEGF-D
Description: VEGF-D values represent serum VEGF-D levels in pg/ml. Higher levels of VEGF-D are associated with Lymphangioleiomyomatosis. A serum VEGF-D greater than 400 pg/ml is a diagnostic biomarker for LAM.
Time Frame: twelve months
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 8 | 7
pg/ml | 572 [294 to 1816] | 944 [350 to 1598]
Statistical Analysis 1: Comparison: Letrozole vs Placebo; Test type: Superiority; p = 0.015, Mixed Models Analysis; Linear Mixed-Effects Model Adjusted for Sirolimus Use. P value was obtained for testing zero slope for log(VEGF-D)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse effects were tabulated using the National Cancer Institute's Common Terminology Criteria for Adverse Events version 4.
Arm/Group | Letrozole | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/8
Other Adverse Events (participants affected / at risk) | 1/9 | 1/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letrozole (N=9) | Placebo (N=8)
worsening dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) — The patient had worsening dyspnea that required hospital admission and resolved slowly without an explanation for the prolonged exacerbation.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letrozole (N=9) | Placebo (N=8)
Swollen lymph nodes (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Endocrine disorder (Endocrine disorders) | 1 (1) | 0 (0)
Blurry vision (Eye disorders) | 1 (1) | 1 (1)
abdominal pain; nausea (Gastrointestinal disorders) | 1 (4) | 1 (10)

LIMITATIONS AND CAVEATS:
Under enrollment. Post menopause not originally assessed by estradiol levels. Small sample sizes led to some imbalances in baseline parameters, such as VEGF-D levels and bronchodilator responsiveness, which could have biased outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No